CLINICAL TRIAL: NCT05518123
Title: A Phase 4, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Tolerability of Rimegepant for the Prevention of Migraine in Adults With a History of Inadequate Response to Oral Preventive Medications
Brief Title: Efficacy and Tolerability of Rimegepant for the Prevention of Migraine in Adults With History of Inadequate Response to Oral Preventive Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BHV3000-407; C4951012 (Other: Alias Study Number); BHV3000-407 (Registry Identifier: CTIS (EU)); 2022-001176-34 (Registry Identifier: CTIS (EU)); 2024-513270-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: Migraine Prevention; Headache; Headache Prevention; Migraine Prevention in adults with inadequate response to oral preventative medications
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rimegepant 75 mg (Experimental)
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75 mg Oral Disintegrating Tablet (ODT) taken every other day during Double-blind Treatment (DBT) phase
  Arms: Rimegepant 75 mg
Drug: Placebo — Matching placebo with every other day dosing during DBT phase
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the efficacy and tolerability of rimegepant for migraine prophylaxis in adults with a history of inadequate response to oral preventive medications

ELIGIBILITY:
Inclusion Criteria:

1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age.
2. Migraine attacks, on average, lasting about 4 - 72 hours, if untreated.
3. 4 to 14 migraine days per month, on average, across the 3 months prior to the Screening Visit (month is defined as 28-days for the purpose of this protocol).
4. Less than15 headache days (migraine or non-migraine) per month in each of the 3-months prior to the Screening Visit and throughout the Screening Phase.
5. Subjects must be able to distinguish migraine attacks from tension/cluster headaches. Prior inadequate response, within 10 years of the Screening Visit, to agents across 2-4 categories of recognized, orally-administered, migraine-preventive medications where at least one example of prior inadequate response is due to lack of efficacy or prior intolerance (not contraindication).

Exclusion Criteria:

1. History of cluster headaches, basilar migraine (migraine with brainstem aura), or hemiplegic migraine.
2. Current medication overuse headaches.
3. 15 or more headache days (migraine or non-migraine) per month in any of the 3-months prior to the Screening Visit or during the first 28- days of the Observation Phase.
4. Inadequate response (due to lack of efficacy, prior intolerance, or contraindication) to agents across > 4 categories of recognized, orally administered, migraine-preventive medications.
5. Active chronic pain syndrome (such as fibromyalgia, chronic pelvic pain, complex regional pain syndrome [CRPS]).
6. Other pain syndromes (including trigeminal neuralgia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, interfere with study assessments of safety or efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of rimegepant (75 mg) to placebo | Week 1 to 12 of DBT Phase
  Subjects are dosed every other day, for the preventative treatment of migraine as measured by mean change in number of migraine days per month (28 days) over 12 week DBT Phase. A migraine day is any calendar day in which the subject experiences a qualified migraine headache. This includes any calendar day in which the subject takes an acute migraine-specific medication.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (111):
- United States (23):
  - Clinical Research Institute, Los Angeles, California
  - California Neuroscience Research, LLC, Sherman Oaks, California
  - Ki Health Partners LLC, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Sandhill Research, LLC d/b/a Accel Research Sites Network-Edgewater Clinical Research Unit, Edgewater, Florida
  - Wr-Msra,Llc, Lake City, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites Network - Ormond Clinical Research Unit, Ormond Beach, Florida
  - Boston Clinical Trials, Boston, Massachusetts
  - Community Clinical Research Network, Inc., Marlborough, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Rochester Medical Group, Rochester Hills, Michigan
  - Clinvest Research, LLC, Springfield, Missouri
  - St Charles Clinical Research, Weldon Spring, Missouri
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Albuquerque Clinical Trials. Inc., Albuquerque, New Mexico
  - DiGiovanna Institute for Medical Education And Research, North Massapequa, New York
  - Headache Wellness Center, PC, Greensboro, North Carolina
  - Synexus Clinical Research US, Inc. - Anderson, Anderson, South Carolina
  - Alliance for Multispecialty Reseach, LLC, Knoxville, Tennessee
  - Red Star Research, LLC, Lake Jackson, Texas
  - DM Clinical Research, Tomball, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- USC Clinical Trials Sunshine Coast, Sippy Downs, Queensland, Australia
- Austria (2):
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
- Belgium (6):
  - UZ Brussel, Jette, Brussels Capital
  - GZA Ziekenhuizen, Antwerp
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Jessa Ziekenhuis, Hasselt
  - Clinique de la Citadelle, Liège
  - Cabinet Privé Dr. Simona Sava, Saint Nicolas Province de Liège
- Canada (5):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - NeuPath Centre for Pain and Spine, Brampton, Ontario
  - Centre de Recherche Saint-Louis/Clinique Neuro-Levis, Lévis, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - ALPHA Recherche Clinique, Québec
- Denmark (4):
  - Bispebjerg Hospital, Copenhagen NV, Capital Region
  - Danish Headache Center, Glostrup Municipality, Capital Region
  - University Hospital of Southern Denmark, Esbjerg
  - Hospitalsenhed Midt, Viborg
- Finland (3):
  - Terveystalo Ruoholahti, Helsinki, Uusimaa
  - Terveystalo Tampere, Tampere
  - Terveystalo Pulssi, Turku
- Germany (9):
  - Schmerz- und Palliativzentrum Göppingen, Göppingen, Baden-Wurttemberg
  - Zentrum für klinische Forschung, Bad Homburg, Hesse
  - Synexus Clinical Research GmbH Synexus Frankfurt Clinical Research Centre, Frankfurt am Main, Hesse
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main, Hesse
  - Intermed GmbH, Wiesbaden, Hesse
  - Studienzentrum Nordwest, Westerstede, Lower Saxony
  - Synexus - Prüfzentrum Leipzig, Leipzig, Saxony
  - Synexus - Prüfzentrum Berlin, Berlin
  - Neuropoint GmbH, Ulm Baden-Wuerttemberg
- Italy (7):
  - IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, MI
  - AOU Luigi Vanvitelli, Napoli, Naples
  - IRCCS San Raffaele, Rome, Rome/lazio
  - SOD Centro Cefalee e Farmacologia Clinica, AOU Careggi, Florence
  - IRCCS Fondazione Besta, Milan
  - University Modena e Reggio Emilia, Modena
- Mexico (6):
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli, State of Mexico
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Medical Care and Research S.A. de C.V., Mérida, Yucatán
  - Centro de Investigación Médica de Aguascalientes (CIMA), Aguascalientes
  - Clinstile, SA de CV, Mexico City
  - Operadora Unidad de Investigación En Salud de Chihuahua, Sa de Cv, Mexico City
- Poland (15):
  - Centrum Medyczne Neuromed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól, Lubusz Voivodeship
  - Centermed Kraków Sp. Z o.o., Krakow, Malopolska
  - Concept Medica, Warsaw, Masovian Voivodeship
  - Dr Sekowska Leczenie Bolu, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Damiana Walbrzyska, Warsaw, Masovian Voivodeship
  - Instytut Zdrowia, Oświęcim, Małopolska
  - Centrum Medyczne Pratia Katowice, Katowice
  - Vita Longa Sp. Z o.o., Katowice
  - MICS Centrum Medyczne Szczecin, Szczecin
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Premium Clinic Wrocław, Wroclaw
  - Centrum Medyczne OPOROW, Wroclaw
  - Centrum Leczenia Bolu dr n med Lukasz Kmieciak, Lodz, Łódź Voivodeship
- Spain (14):
  - Hospital Universitario de Elda, Elda, Alicante
  - Hospital Clinic de Barcelona Plato Headquarters, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Ruber Juan Bravo, Salamanca
  - University Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Virgen del Rocio University Hospital, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Consorcio Hospital General Universitario, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Sweden (7):
  - CTC Solna, Solna, Stockholms LÄN [se-01]
  - CTC MTC, Uppsala, Uppsala LÄN [se-03]
  - Carlanderska Hospital, Gothenburg
  - Skåneuro Privatmottagning, Lund
  - Hälsoklustret, Stockholm
  - Akardo Med Site, Stockholm
  - University Hospital Uppsala (VO Neuro), Uppsala
- United Kingdom (9):
  - Re: Cognition Health Ltd., Edgebaston, Birmingham
  - Hull University Hospitals NHS Trust, Hull, EAST Riding
  - 4 Medical Clinical Solutions London, Ilford, Essex
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - Lakeside Healthcare Group Research, Corby, Northamptonshire
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Cognition Health - Bristol, Bristol
  - Kings College London, London
  - 4 Medical Clinical Solutions, Swinton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Pozo-Rosich P, Lopez JAG, Lisewski P, Aslan AN, Seehra H, Thiry A, Abraham L, Ramirez LM, Fountaine R, Fullerton T. A phase 4, randomized, double-blind, placebo-controlled trial evaluating the efficacy and tolerability of rimegepant for the prevention of episodic migraine in adults with a history of inadequate response to traditional oral preventive medications. Cephalalgia. 2025 Nov;45(11):3331024251391378. doi: 10.1177/03331024251391378. Epub 2025 Nov 18. PMID 41255098
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-407